CLINICAL TRIAL: NCT01852643
Title: Determine and Compare the Finding of Rhinomanometry Before and After Treatment in Two Ways of Rhinoplasty Surgery (Spreader Graft and Lateral Crural Over Lapping)
Brief Title: Spreader Graft and Lateral Crural Overlay Technique in Rhinoplasty
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Amiryousef Ahmadnia, Dr., Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 390548
Record Dates: First submitted 2013-05-09; First posted 2013-05-14 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Rhinoplasty Techniques
Keywords: Rhinoplasty; Spreader graft technique; Lateral crural overlay technique; Rhinomanometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spreader graft (Active Comparator)
  Interventions: Procedure: Spreader graft
- Lateral crural overlay (Active Comparator)
  Interventions: Procedure: Lateral crural overlay

INTERVENTIONS:
Procedure: Spreader graft — Spreader graft technique is performed by a group of expert surgeons.
  Arms: Spreader graft
Procedure: Lateral crural overlay — Lateral crural overlay technique is performed by a group of expert surgeons.
  Arms: Lateral crural overlay

SUMMARY:
Most of the studies performed to compare the present techniques of rhinoplasty have been based on the clinical examination and change of postoperative complaints that cannot be very precise in evaluating the advantages of one technique over another. Therefore, in this study the investigators are going to compare the efficacy of spreader graft and lateral crural overlay techniques by an objective method, rhinomanometry.

ELIGIBILITY:
Inclusion Criteria:

* Candidates of rhinoplasty
* Willingness to participate

Exclusion Criteria:

* Having structural problems such as nasal obstruction
* History of the deformity requiring rhinoplasty of the deviated septum
* Hardening surgery
* New clinical conditions or a change in therapeutic technique
* Unwillingness to continue participating in the study
* Having no access to subjects after the operation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Nasal flow | Up to 3 months
  Rhinomanometry is performed by a technician in two stages: before surgery and three months after surgery. It is performed in line with the standards suggested by the "Committee Report on Standardization of Rhinomanometry". After surgery, patients are monitored for one month and rhinomanometry is performed under the same initial conditions after three months. In both stages of rhinomanometry, nasal resistance means are evaluated by Pascal per milliliter per second (Pa/mL/s) and the right and left and total nasal flow indices are evaluated by milliliter per second (mL/s).
Nasal resistance | Up to 3 months
  Rhinomanometry is performed by a technician in two stages: before surgery and three months after surgery. It is performed in line with the standards suggested by the "Committee Report on Standardization of Rhinomanometry". After surgery, patients are monitored for one month and rhinomanometry is performed under the same initial conditions after three months. In both stages of rhinomanometry, nasal resistance means are evaluated by Pascal per milliliter per second (Pa/mL/s) and the right and left and total nasal flow indices are evaluated by milliliter per second (mL/s).

CONTACTS AND LOCATIONS:
Overall Officials: Amiryousef Ahmadnia, MD, Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Department of Plastic Surgery, Alzahra Hospital, Isfahan, Isfahan, Iran